CLINICAL TRIAL: NCT02273934
Title: The Effectiveness of Reablement in Home Dwelling Adults. A Quasi Experimental Trial
Brief Title: The Effectiveness of Reablement in Home Dwelling Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Frode F. Jacobsen (Other)
Collaborators: University of Oslo (Other); University of Bergen (Other)
Responsible Party: Sponsor-Investigator, Frode F. Jacobsen, Professor, Bergen University College
Organization: Bergen University College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EL-123-REHAB
Record Dates: First submitted 2014-09-29; First posted 2014-10-24 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-06

CONDITIONS: Physical Disability
Keywords: Home-based rehabilitation; Activities of daily living; Restorative care; Reablement; Everyday rehabilitation
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reablement (Experimental): Reablement is an intensive, multidisciplinary, client-centered, home-based type of rehabilitation, where ordinary activities of daily living are used for rehabilitative purposes. It is a rehabilitation alternative that may be offered to adults, and there is no lower age limit. An occupational therapist and physical therapist, or nurse, constitutes the key personal, while home helpers, assistants and others with lower education, are the ones who work rehabilitative with the person on a daily basis focusing on self-help.
  Interventions: Behavioral: Reablement
- Standard treatment (Active Comparator): This arm consists of the standard treatment home-dwelling elderly persons receive when applying for home-based help. Some elderly may receive home-based nursing or home help services assisting them in daily activities, while others may receive occupational therapy or physical therapy measures for rehabilitative purposes.
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Reablement — The intervention deals with improving function in daily activities the person defines as important in the areas of self-care, productivity and leisure.
  Other Names: Hverdagsrehabilitering; Hemrehabilitering; Re-ablement; Restorative care
  Arms: Reablement
Behavioral: Standard treatment — The control intervention is standard home-based treatment/care in Norway.
  Other Names: Usual care; Treatment as usual
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to determine whether a special kind of rehabilitation offered to home-dwelling adults is effective with regards to functional ability, health-related quality of life, coping, mental health and municipal costs.

DETAILED DESCRIPTION:
Health promotion and prevention of functional decline among home dwelling adults and immediate onset of rehabilitation, can improve function, and reduce or delay need for home-based assistance and institution placement. In the coming years there will be a significant increase in number of persons in Norway that need interventions aiming at coping with everyday activities. Therefore there is a call for new models for early intervention and rehabilitation in order to give service to a larger amount of home living people. Reablement is a new and promising rehabilitation model which many Norwegian municipalities are implementing in order to meet current and future needs for municipal home-based services. However, very little research has been performed regarding the effectiveness of this intervention. This study aims at assessing the effectiveness of reablement in terms of daily functioning, health-related quality of life, coping, mental health and economic municipal costs.

The study will be conducted in 44 municipalities in Norway. It is a quasi-experimental intervention trial, recruiting home-dwelling adults with an initial functional decline in daily activities. The intervention is intensive, multidisciplinary, home-based rehabilitation given by home-trainers, under supervision from an occupational therapist, nurse or a physiotherapist. The control intervention is standard home-based treatment and care.

A total of approximately 750 participants will be recruited, including approximately 100 participants the control group. The participants will be assessed at baseline, and at 10 weeks ,6-, and 12 months follow-up. Primary outcomes will be participation, activity, and municipal expenditures. Costs are generated by the working hours of the different professions. Hence, there will be a weekly registration of the working hours different health care professions spend in the private homes of the participants.

Data analyses will be performed according to intention to treat. Univariate analysis of covariance will be used to investigate differences between the groups from baseline to the end of intervention. The working hour data is panel data and will be analyzed accordingly; a random or a mixed effect regression model will be employed. Also, descriptive statistics and simpler tests will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Home-dwelling person
* Applicant of home-based services
* Above 18 years old
* Functional decline in at least one activity
* Able to understand written and oral Norwegian

Exclusion Criteria:

* Cognitive disability
* Terminal ill
* Being assessed as needing nursing home placement
* Being assessed as needing institution-based rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in score in Canadian Occupational Performance Measure | Baseline, 10 weeks, 6 months and 12 months
  Activity and participation will be measured using Canadian Occupational Performance Measure (COPM) The COPM is a measure of a client's self-perception of occupational performance in the areas of self-care, productivity and leisure. Outcome measures for the COPM are: the client's most important problems in occupational performance and a total score of performance and a total score of satisfaction for these problems.

SECONDARY OUTCOMES:
Expenditure | Weekly from baseline to 6 months
  Municipal expenditures will be recorded weekly for six months. Costs will be recorded in accordance with the operating hours of the different health care professions in the private homes of the participants.
Short Physical Performance Battery | Baseline, 10 weeks, 6 months and 12 months
  Short Physical Performance Battery (SPPB) investigates balance, walking function and muscle strength in the lower limbs.

OTHER OUTCOMES:
Health-related Quality of Life | Baseline, 10 weeks, 6 months and 12 months
  Health-related Quality of Life (EQ-5D) measures health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses.
Sense of coherence | Baseline, 10 weeks, 6 months and 12 months
  Sense of coherence (SOC) measures comprehensibility (5 items), manageability (4 items) and meaning (4 items).
Mental Health Continuum | Baseline, 10 weeks, 6 months and 12 months
  Mental Health Continuum Short Form (MHC-SF) measures emotional (3 items), psychological (6 items) and social (5 items) well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Frode Jacobsen, PhD, Study Chair — Bergen University College
Locations (1):
- Bergen University College, Bergen, Bergen, Norway

REFERENCES:
- [Derived] Langeland E, Tuntland H, Folkestad B, Forland O, Jacobsen FF, Kjeken I. A multicenter investigation of reablement in Norway: a clinical controlled trial. BMC Geriatr. 2019 Jan 30;19(1):29. doi: 10.1186/s12877-019-1038-x. PMID 30700255
- [Derived] Langeland E, Tuntland H, Forland O, Aas E, Folkestad B, Jacobsen FF, Kjeken I. Study protocol for a multicenter investigation of reablement in Norway. BMC Geriatr. 2015 Sep 15;15:111. doi: 10.1186/s12877-015-0108-y. PMID 26374305
- See also: Published study protocol — https://www.researchgate.net/publication/281938720_Erratum_to_Study_protocol_for_a_multicenter_investigation_of_reablement_in_Norway